CLINICAL TRIAL: NCT04750616
Title: NAD+ Augmentation in Cardiac Surgery Associated Myocardial Injury (NACAM) Trial
Brief Title: NAD+ Augmentation in Cardiac Surgery Associated Myocardial Injury Trial
Acronym: NACAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Beth Israel Deaconess Medical Center (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1620125
Record Dates: First submitted 2021-01-29; First posted 2021-02-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Ischemia Reperfusion Injury; Myocardial Injury; Acute Kidney Injury
MeSH Terms: conditions — Reperfusion Injury; Acute Kidney Injury | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral niacinamide (Experimental)
  Interventions: Drug: Niacinamide
- Matched placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niacinamide — Niacinamide 3 grams on the day of surgery and post-surgical days one and two
  Arms: Oral niacinamide
Drug: Placebo — Matched placebo on the day of surgery and post-surgical days one and two
  Arms: Matched placebo

SUMMARY:
A Randomized, Double-blind, placebo-controlled Trial to Evaluate the Efficacy of Oral Nam for the Prevention of Acute Kidney Injury in Patients Undergoing On-Pump Cardiac Surgery

DETAILED DESCRIPTION:
This trial is a single-center, randomized, double-blind placebo-controlled Trial of Nam versus placebo in patients undergoing on-pump cardiac surgery. After screening and enrollment, patients will be stratified according to CKD status (eGFR<45 ml/min/m2) and surgical site and randomized in a 1:1 manner to receive either Nam 3 grams or placebo on the day of surgery and post-surgical days one and two.

The overall trial duration is planned for 42 months, consisting of 39 months of active recruitment and treatment period and three months of follow-up from the last patient enrolled.

ELIGIBILITY:
Inclusion Criteria

* Informed consent before any study-related activities.
* Men or women >18 years of age who are scheduled for non-emergent cardiac surgery procedures requiring CPB and are at increased risk for surgery-related adverse cardiovascular outcomes.

Procedures include:

* CABG
* Aortic, mitral, tricuspid, or pulmonic valve replacement or repair
* CABG with aortic, mitral, tricuspid, and/or pulmonic valve replacement

Risk factors for surgery related to adverse cardiovascular outcomes include one or more of the following:

* Valve surgery
* eGFR < 45 ml/min/1.73m2
* Documented LVEF ≤ 35% within six months before surgery
* Documented history of heart failure
* Insulin-requiring diabetes
* Non-insulin-requiring diabetes and the presence of ≥+2 proteinuria on urinalysis (or equivalent on urine protein-to-creatinine ratio or urine albumin-to-creatinine ratio)
* Preoperative anemia (hemoglobin <11g/dl for men and women)
* History of prior CABG
* Age ≥65

Exclusion Criteria

* Preexisting AKI within seven days before surgery as defined by KDIGO stage ≥1 (serum creatinine-based)
* Kidney transplant status
* Off-pump cardiac surgery
* ESRD
* Emergent cardiac surgery
* Pregnancy
* Patient enrolled in competing research studies that may affect outcomes
* Patients held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Troponin T AUC | From baseline to three days after surgery
  Troponin T AUC, composed of single daily serum measurements

SECONDARY OUTCOMES:
Mean difference in uQuin/Tryp ratio AUC | From baseline to three days after surgery
  Mean difference in uQuin/Tryp ratio AUC composed of single daily serum measurements
Mean difference in eGFR | From baseline through day 5.
  Mean difference in eGFR (CKD-EPI formula)

OTHER OUTCOMES:
Number of Participants with the following Adverse Events and Serious Adverse Events | From baseline through day 90
  * Postoperative dysrhythmias
  * Postoperative re-hospitalization.
  * Heart failure
  * Surgical wound infection
  * Transfusion requiring perioperative bleed
  * Post-surgical deep vein thrombosis and pulmonary emboli
  * Nosocomial infection
  * Nausea and vomiting
  * Adverse events leading to treatment discontinuation
  * Perioperative liver injury (x2 upper normal-limit)
  * Post-operative thrombosis and pulmonary emboli
  * Impairment of renal function (KDIGO AKI)
Length of index hospital stay. | From baseline through day 90
  • Mean length of index hospital stay (days)
Length of intensive care unit stay. | From baseline through day 90
  • Mean length of intensive care unit stay (days)
Perioperative inotropic-score and vasoactive-inotropic score. | At 6, 12, 24, and 48 hours post operatively
  • Mean inotropic-score and vasoactive-inotropic score
Perioperative fluid volume administration. | From baseline through day 2
  • Mean daily perioperative fluid volume administration
Perioperative brain-natriuretic peptide AUC | From baseline to three days after surgery
  BNP AUC, composed of single daily serum measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente San Francisco Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scurt FG, Bose K, Mertens PR, Chatzikyrkou C, Herzog C. Cardiac Surgery-Associated Acute Kidney Injury. Kidney360. 2024 Jun 1;5(6):909-926. doi: 10.34067/KID.0000000000000466. Epub 2024 May 1. PMID 38689404